CLINICAL TRIAL: NCT06894706
Title: Lanzhou Anning District People's Hospital
Brief Title: The Impact of Functional Exercise Training on Postoperative Knee Joint Recovery in Patients with Meniscal Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biao Yang (Other Government)
Responsible Party: Sponsor-Investigator, Biao Yang, Lanzhou Anning District People's Hospital, Lanzhou Anning District People's Hospital
Organization: Lanzhou Anning District People's Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: No. 20240927
Record Dates: First submitted 2025-03-10; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-09

CONDITIONS: Functional Exercise Training; Knee Meniscus Injury; Knee Joint Function
Keywords: Functional exercise training; knee meniscus injury; knee joint function
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control （CON） group (Other): Both groups were given arthroscopy and meniscoplasty. After operation, the control group received active knee flexion and extension exercise, ankle pump training, quadriceps muscle training and other routine rehabilitation training.
  Interventions: Behavioral: Control （CON） group
- Functional exercise training (FET) group (Other): Patients in the observation group were supplemented with neuromuscular training on the basis of routine rehabilitation training, and received rehabilitation education before training. The patients were informed of the specific content, frequency, expected effect and importance of training in various forms such as on-site demonstration combined with publicity brochures and playing videos, so as to improve patient cooperation.
  Interventions: Behavioral: Functional exercise training (FET) group

INTERVENTIONS:
Behavioral: Control （CON） group — Both groups were given arthroscopy and meniscoplasty. After operation, the control group received active knee flexion and extension exercise, ankle pump training, quadriceps muscle training and other routine rehabilitation training.
  Arms: Control （CON） group
Behavioral: Functional exercise training (FET) group — Patients in the observation group were supplemented with neuromuscular training on the basis of routine rehabilitation training, and received rehabilitation education before training. The patients were informed of the specific content, frequency, expected effect and importance of training in various forms such as on-site demonstration combined with publicity brochures and playing videos, so as to improve patient cooperation.
  Arms: Functional exercise training (FET) group

SUMMARY:
AIM: To investigate the impact of functional exercise training on postoperative functional recovery in patients with knee meniscus injuries.

METHODS:A prospective randomized controlled trial (RCT) was conducted from April 2023 to September 2024, involving 96 patients with knee meniscus injuries who underwent meniscus repair interventions. Participants were randomly assigned to either the Control （CON） group (n=48) or the functional exercise training (FET) group (n=48) using a computer-generated random number table. The CON group received standard rehabilitation, while the FET group underwent functional exercise training. Clinical outcomes were evaluated at baseline, 1 month, and 6 months post-intervention, including the Lysholm score, IKDC score, VAS pain score, range of motion (ROM), serum levels of prostaglandin E2 (PGE2) and serotonin (5-HT), as well as passive 60° position sense and 60° motion sense. Postoperative complications occurring within 1 month were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* meniscus injury was diagnosed by magnetic resonance imaging; meniscoplasty was performed; No shedding occurred during follow-up.

Exclusion Criteria:

* Patients with joint dislocation and fracture; poor compliance; severe osteoarthritis, rheumatoid arthritis; Combined with metabolic diseases, coagulation disorders and serious organic diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Demographic data comparison | baseline, pre-intervention

SECONDARY OUTCOMES:
Lysholm Knee Scoring Scale scores | up to 24 weeks
  The Lysholm Knee Scale (Lysholm Knee Scale) is a widely used assessment tool to measure the functional status and quality of life of the knee joint, especially in the assessment of recovery after knee injury and surgery. The scale quantifies knee function through eight items (such as claudication, pain, stability, etc.), with a total score ranging from 0 to 100, with higher scores indicating better knee function. The Lysholm Scale is designed to provide clinicians with an effective assessment tool to help them judge the impact of knee disease and injury. The MCID is 10 points.
International Society of Knee Injuries and Arthroscopy Score | up to 24 weeks
  IKDC (International Knee Injury and Arthroscopy Score) is a tool used to assess knee function and symptoms and is widely used in rehabilitation assessment of knee injuries, especially in recovery monitoring after anterior cruciate ligament and meniscus injuries. The rating scale includes four main items: symptoms (pain, swelling, etc.), activity (functional limitations in daily activities), motor capacity (performance in physical activities), and function (knee stability and load-bearing capacity). The IKDC score is scored on a scale of 0 to 100, with 0 indicating complete loss of knee function and 100 indicating complete recovery and normal function of the knee. The higher the score, the better, indicating better knee function and less severe symptoms. The MCID (minimum clinically significant difference) of IKDC is usually 10 points.
Range of Motion | up to 24 weeks
Visual Analog Scale | up to 24 weeks
  Visual analog scale (VAS) is a commonly used subjective pain assessment tool, which is widely used in clinical practice and research. It is usually scored on a scale of 0 to 10, which is explained as follows: 0: completely painless. 1 to 3 points: mild pain, does not affect daily life. Scores 4 to 6: Moderate pain that interferes with daily activities and sleep. Score 7 to 10: Severe pain that severely affects quality of life and daily functioning. MCID is usually 2 points.
Passive position sense | up to 24 weeks
  The sensory threshold measurement method was used to measure passive position perception, motion perception and isotonic power. During the passive 60° position perception test, subjects were asked to sit and stop when they felt reaching the target Angle with an eye mask and headset. Each Angle was repeated three times. Record the error between the target Angle and the measured Angle; 10% of the maximum contraction force of the quadriceps isometric resistance was selected, and the activity Angle of the knee joint was set as the activity degree of the knee joint in the seated position. 60 was measured on a CPM machine using a motion test sensor. The subjects passively completed 60° knee flexion and extension at a constant angular speed of 1° / s. The subjects stopped the movement when they felt the joint movement or the joint position change. Three tests were conducted and the Angle of each perceived movement was recorded.
Kinesthesia test | up to 24 weeks
Prostaglandin E2 | up to 24 weeks
5-hydroxytryptamine | up to 24 weeks
complications | up to 24 weeks
  The incidence of complications in the first month after operation was measured

CONTACTS AND LOCATIONS:
Locations (1):
- Lanzhou Anning District People's Hospital, Lanzhou, China

IPD SHARING:
Plan to Share IPD: No